CLINICAL TRIAL: NCT05059067
Title: Macintosh Blade Size During Laryngoscopy for Endotracheal Intubation. A Prospective Observational Study.
Acronym: MacSize
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 00010254-2021-016
Record Dates: First submitted 2021-06-15; First posted 2021-09-28 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-06

CONDITIONS: Endotracheal Intubation
Keywords: Intubation; Macintosh blade; Laryngoscopie; Operative room; Intensive Care Unit; Emergency department
MeSH Terms: conditions — Emergencies | interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Macintosh blade size 3: Patients intubated using Macintosh blade size 3
  Interventions: Device: Direct laryngoscopy for endotracheal intubation
- Macintosh blade size 4: Patients intubated using Macintosh blade size 4
  Interventions: Device: Direct laryngoscopy for endotracheal intubation

INTERVENTIONS:
Device: Direct laryngoscopy for endotracheal intubation — Patients in operative room, intensive care unit and emergency department requiring direct laryngoscopy for endotracheal intubation

SUMMARY:
Endotracheal intubation is a frequent procedure in the operating room, in intensive care units and in emergency medicine (in- or out-of-hospital) but optimal Macintosh blade size remains unknown to date.

DETAILED DESCRIPTION:
Endotracheal intubation is an extremely frequent procedure in the operating room, in intensive care units and in emergency medicine (in- or out-of-hospital). Apart from special cases of foreseen difficult programmed intubation, direct laryngoscopy remains the most frequently used technique. It requires the use of a handle (short or long), which serves as a light source on which is adapted a Macintosh curved blade, metallic or plastic, single or multiple use. The choice of blade size is based on the experience of the physician. Most often, in adult settings, size 3 or 4 blades are used. The very spartan literature on the subject and the current recommendations do not provide any information on the choice of blade size. We therefore wish to evaluate these practices in terms of success of the first laryngoscopy, Cormack-Lehane and POGO (percentage of glottic opening visualized) scores, the need to use an alternative technique or a second operator. The results will be analyzed with regard as a function and experience of the person performing the laryngoscopy, as well as the setting (urgent or scheduled). These data are usually collected during the performance of an endotracheal intubation whatever the circumstances: operating room, intensive care unit and emergency department (in-hospital) and in the SAMU-SMUR (pre-hospiatl medical service) at Clermont-Ferrand University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be admitted in an operative room, an intensive care unit (ICU) or an emergency department and require mechanical ventilation through an orotracheal tube.
* Adult (age ≥ 18 years)
* Subjects must be covered by public health insurance
* Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency.

Exclusion Criteria:

* Anticipated difficult intubation requiring videolaryngoscopy
* Nasotracheal intubation
* Refusal of study participation or to pursue the study by the patient
* Absence of coverage by the French statutory healthcare insurance system
* Protected person

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient requiring orotracheal intubation with direct laryngoscopy
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with successful first-pass orotracheal intubation | At intubation
  The proportion of patients with successful first-pass orotracheal intubation

SECONDARY OUTCOMES:
Severe complications related to intubation_hypoxemia | At intubation
  Rate of severe hypoxemia defined by lowest oxygen saturation (SpO2) < 80 %
Severe complications related to intubation_severe collapse | At intubation
  Rate of cardiovascular collapse, defined as systolic blood pressure less than 65 mm Hg recorded at least once or less than 90 mm Hg lasting 30 minutes despite 500-1,000 ml of fluid loading (crystalloids solutions) or requiring introduction or increasing doses by more than 30% of vasoactive support
Severe complications related to intubation_cardiac arrest | At intubation
  Rate of cardiac arrest
Severe complications related to intubation_death | At intubation
  Rate of death during intubation
Moderate complications related to intubation_difficult intubation | At intubation
  Rate of difficult intubation
Moderate complications related to intubation_arrythmia | At intubation
  Rate of severe ventricular or supraventricular arrhythmia requiring intervention
Moderate complications related to intubation_oesophageal intubation | At intubation
  Rate of oesophageal intubation
Moderate complications related to intubation_agitation | At intubation
  Rate of agitation
Moderate complications related to intubation_aspiration | At intubation
  Rate of pulmonary aspiration
Moderate complications related to intubation_dental injuries | At intubation
  Rate of dental injuries
Cormack Lehane | During intubation
  Rate of Cormack-Lehane grade of glottic view
Difficulty of intubation | During intubation
  Rate of operator-assessed difficulty of intubation
Additional airway equipment | During intubation
  Rate of need for additional airway equipment (video laryngoscope, bougie, stylet, fibroscope, cricothyrotomy)
Additional second operator | During intubation
  Rate of need for a second operator
POGO (percentage of glottic opening) | During intubation
  Rate of POGO grade of glottic view

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Godet, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France